CLINICAL TRIAL: NCT02566044
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of Inhaled QBW276 in Patients With Cystic Fibrosis
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics Study of Inhaled QBW276 in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CQBW276X2201; 2014-004915-35 (EudraCT Number)
Record Dates: First submitted 2015-09-18; First posted 2015-10-01 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2019-06

CONDITIONS: Pulmonary Cystic Fibrosis
Keywords: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CQBW276 (Experimental): Cohorts 1 and 2 will enroll 8 patients each (6:2 QBW276 and placebo, respectively).
  Cohort 1: dose is 3 mg bid (6 mg daily) QBW276 or placebo for 7 days. Cohort 2: dose and frequency will be confirmed after cohort 1 is complete. The duration is 14 days.
  Cohort 3: dose and frequency will be confirmed after cohort 2 is complete. The duration is approximately 4 months. Patients will be randomized to one of two treatment sequences: QBW276 in Period 1 and Placebo in Period 2 or Placebo in Period 1 and QBW276 in Period 2. Twenty four patients are required to complete cohort 3.
  Interventions: Drug: QBW276
- Placebo (Placebo Comparator): Cohorts 1 and 2 will enroll 8 patients each (6:2 QBW276 and placebo, respectively).
  Cohort 1: dose is 3 mg bid (6 mg daily) QBW276 or placebo for 7 days. Cohort 2: dose and frequency will be confirmed after cohort 1 is complete. The duration is 14 days.
  Cohort 3: dose and frequency will be confirmed after cohort 2 is complete. The duration is approximately 4 months. Patients will be randomized to one of two treatment sequences: QBW276 in Period 1 and Placebo in Period 2 or Placebo in Period 1 and QBW276 in Period 2. Twenty four patients are required to complete cohort 3.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Placebo
  Arms: Placebo
Drug: QBW276 — 0.3 mg and 1.5 mg strengths
  Arms: CQBW276

SUMMARY:
This is a study of multiple doses of inhaled QBW276 in patients with cystic fibrosis on top of standard of care. The study was divided into 3 Cohorts. Cohorts 1 and 2 are designed to be a randomized, double-blind, placebo-controlled, parallel arm, multiple dose study to assess the safety, tolerability, pharmacokinetics, and preliminary efficacy of inhaled QBW276 over 1 week (cohort 1) or 2 weeks (cohort 2) in patients with cystic fibrosis regardless of their genotype.

The study was terminated after Cohort 2 due to the resource issues.

ELIGIBILITY:
Inclusion Criteria:

* Cohorts 1 and 2 = any genotype on any standard of care treatment
* Cohort 3 = F508del homozygotes on standard of care at that time
* FEV₁between 40 and 100%
* LCI2.5 ≥ 8 if FEV₁is more than 80%

Exclusion Criteria:

* Adrenal or electrolyte abnormalities
* Lung transplant
* Autonomic dysfunction (e.g. recurrent episodes of fainting, palpitations, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (2):
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Dallas, Texas
- Germany (2):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Essen

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=280

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated after completion of all randomized patients in Cohort 2 due to strategic issues. All patients completed the study prior to termination.
Groups:
- Cohort 1 QBW276: QBW276 3mg bid
- Cohort 2 QBW276: QBW276 6mg bid
- Placebo: Placebo to QBW276 dose 3mg bid Cohort 1, and Placebo to QBW276 dose 6mg bid Cohort 2.
Period: Overall Study
Arm/Group | Cohort 1 QBW276 | Cohort 2 QBW276 | Placebo
Started | 6 | 6 | 4
Completed | 6 | 6 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 QBW276 | Cohort 2 QBW276 | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.5 (7.66) | 34.8 (8.06) | 28.8 (11.53) | 33.9 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 0 | 3
  Male | 6 | 3 | 4 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 6 | 4 | 16
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cohorts 1 and 2: Safety Assessments, Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]).
Description: Adverse events were summarized by the number of patients having any adverse event overall and presented in the safety section. Study was prematurely terminated
Time Frame: Cohort 1: day 1-7; Cohort 2: day 1-14
Population: Safety set: The safety analysis set included all patients that received any study drug
Measure: Number; unit: Participants
Arm/Group | Cohort 1 QBW276 | Cohort 2 QBW276 | Placebo
Number analyzed (Participants) | 6 | 6 | 4
Participants
  Death | 0 | 0 | 0
  Serious AE | 0 | 0 | 0
  Subjects with at least one AE | 2 | 6 | 0

2. Primary Outcome: Cohorts 1 and 2: Pharmacokinetics (Cmax) of QBW276, QBP545, and QBV697 in Plasma
Description: Blood collection will be used to observe the maximum plasma concentration (Cmax) following administration of QBW276. Pharmacokinetic blood samples were collected at the time points. In Cohorts 1 and 2 this consisted of multiple samples through 6 hours after inhalation on Days 1 and 7 in Cohort 1 and Days 1 and 14 in Cohort 2 with predose samples on selected days. The Cmax, was determined using the actual recorded sampling times and noncompartmental methods. Since steady state was likely reached by Day 7, Cmax on Days 7 or 14 correspond to Cmax,ss
Time Frame: Cohort 1: day 1, 7; Cohort 2: day 1, 14
Population: Pharmacokinetic set: The PK analysis set included all patients with at least one available valid (i.e., not flagged for exclusion) PK concentration measurement, who received study drug, and experienced no protocol deviations with relevant impact on PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cohort 1 QBP545; Cohort 2 QBP545: formation of metabolites QBP545
- Cohort 1 QBV697; Cohort 2 QBV697: formation of metabolites QBV697
Arm/Group | Cohort 1 QBW276 | Cohort 1 QBP545 | Cohort 1 QBV697 | Cohort 2 QBW276 | Cohort 2 QBP545 | Cohort 2 QBV697
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng/mL
  Day 1: number analyzed (Participants) | 2 | 6 | 6 | 4 | 6 | 6
  Day 1 | 0.159 (NA) | 3.88 (1.38) | 1.21 (0.415) | 0.174 (0.0716) | 5.98 (3.72) | 1.63 (0.931)
  Day 7: number analyzed (Participants) | 3 | 6 | 6 | 0 | 0 | 0
  Day 7 | 0.145 (0.114) | 5.46 (1.26) | 1.45 (0.504) |  |  |
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 5
  Day 14 |  |  |  | 0.267 (0.109) | 7.80 (4.34) | 3.07 (1.72)

3. Primary Outcome: Cohorts 1 and 2: Pharmacokinetics (Tmax) of QBW276, QBP545, and QBV697 in Plasma
Description: Blood collection will be used to observe the maximum plasma concentration (Tmax) following administration of QBW276. Pharmacokinetic blood samples were collected at the time points. In Cohorts 1 and 2 this consisted of multiple samples through 6 hours after inhalation on Days 1 and 7 in Cohort 1 and Days 1 and 14 in Cohort 2 with predose samples on selected days. The Tmax, was determined using the actual recorded sampling times and noncompartmental methods. Since steady state was likely reached by Day 7, Tmax on Days 7 or 14 correspond to Tmax,ss
Time Frame: Day 1, 7 and 14
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Cohort 1 QBW276 | Cohort 1 QBP545 | Cohort 1 QBV697 | Cohort 2 QBW276 | Cohort 2 QBP545 | Cohort 2 QBV697
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hr
  Day 1: number analyzed (Participants) | 2 | 6 | 6 | 4 | 6 | 6
  Day 1 | 0.183 [0.167 to 0.200] | 0.375 [0.233 to 0.933] | 0.433 [0.233 to 0.500] | 0.250 [0.167 to 0.250] | 0.250 [0.167 to 2.03] | 0.250 [0.167 to 1.03]
  Day 7: number analyzed (Participants) | 3 | 6 | 6 | 0 | 0 | 0
  Day 7 | 0.183 [0.167 to 0.183] | 0.500 [0.250 to 0.967] | 0.375 [0.167 to 2.0] |  |  |
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6
  Day 14 |  |  |  | 0.258 [0.233 to 0.533] | 0.500 [0.267 to 0.533] | 0.500 [0.233 to 0.533]

4. Primary Outcome: Cohorts 1 and 2: Pharmacokinetics (AUCtau) of QBW276, QBP545, and QBV697 in Plasma
Description: Blood collection will be used to observe the maximum plasma concentration (AUCtau) following administration of QBW276. Pharmacokinetic blood samples were collected at the time points. In Cohorts 1 and 2 this consisted of multiple samples through 6 hours after inhalation on Days 1 and 7 in Cohort 1 and Days 1 and 14 in Cohort 2 with predose samples on selected days. The AUCtau, was determined using the actual recorded sampling times and noncompartmental methods. Since steady state was likely reached by Day 7, AUCtau on Days 7 or 14 correspond to AUClast,ss
Time Frame: Day 1, 7 and 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 1 QBW276 | Cohort 1 QBP545 | Cohort 1 QBV697 | Cohort 2 QBW276 | Cohort 2 QBP545 | Cohort 2 QBV697
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hr*ng/mL
  Day 1: number analyzed (Participants) | 2 | 6 | 6 | 4 | 5 | 6
  Day 1 | 0.0332 (NA) — NA- Not achievable | 14.3 (4.09) | 1.35 (0.827) | 0.0634 (0.0473) | 13.9 (6.57) | 1.79 (1.54)
  Day 7: number analyzed (Participants) | 3 | 6 | 6 | 0 | 0 | 0
  Day 7 | 0.0278 (0.0362) | 18 (4.21) | 1.80 (0.797) |  |  |
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 6 | 5 | 5
  Day 14 |  |  |  | 0.0918 (0.0689) | 30.6 (6.59) | 2.94 (1.59)

5. Primary Outcome: Cohorts 1 and 2: Pharmacokinetics Accumulation Ratio (Racc) of QBW276, QBP545, and QBV697 in Plasma
Description: The accumulation ratio (Racc) will be reported using blood samples taken on days 1 -7 in cohort 1 and days 1-14 in cohort 2. Accumulation ratio (Racc) for QBW276 and metabolites was not calculated by PK software for patients where BLOQ values were observed for all blood samples in their PK profile.
Time Frame: Cohort 1: 7 days; Cohort 2: 14 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Cohort 1 QBW276 | Cohort 1 QBP545 | Cohort 1 QBV697 | Cohort 2 QBW276 | Cohort 2 QBP545 | Cohort 2 QBV697
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
Ratio | 1.20 (0.047) | 1.28 (0.122) | 1.84 (0.384) | 1.59 (0.126) | 1.01 (0.714) | 1.74 (0.765)

6. Secondary Outcome: Cohorts 1 and 2: Change From Baseline in Percent Predicted Forced Expiratory Volume in the First Second by Spirometry (% Predicted FEV1)
Description: To evaluate the response to multiple doses of inhaled QBW276 in percent predicted forced expiratory volume in the first second by spirometry according to international standards over 1 or 2 weeks of treatment compared with placebo in patients with cystic fibrosis.
Time Frame: Baseline to End of study (EOS)
Population: Pharmacodynamics analysis set: The PD analysis set included all patients with available PD data and no major protocol deviations with relevant impact on PD data.
Measure: Mean (Standard Deviation); unit: Percent predicted FEV1
Arm/Group | Cohort 1 QBW276 | Cohort 2 QBW276 | Placebo
Number analyzed (Participants) | 6 | 6 | 4
Percent predicted FEV1 | -0.1 (2.30) | -0.1 (1.32) | -2.7 (3.71)

7. Secondary Outcome: Cohorts 1, 2: Change From Baseline in Lung Clearance Index (LCI) From Baseline to Day 7 for Cohort 1, Day 14 for Cohort 2.
Description: Change in Lung Clearance Index (LCI) will be conducted by multiple breath nitrogen washout according to international standards
Time Frame: Baseline to EOS
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1 QBW276 | Cohort 2 QBW276 | Placebo
Number analyzed (Participants) | 6 | 6 | 4
Ratio | 1.530 (2.0167) | 2.478 (3.1397) | 0.470 (0.4101)

ADVERSE EVENTS:
Time Frame: Up to 18 days
Groups:
- Cohort 1 QBW276: QBW276 3 mg bid
- Cohort 2 QBW276: QBW276 6 mg bid
Arm/Group | Cohort 1 QBW276 | Cohort 2 QBW276 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 2/6 | 6/6 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 QBW276 (N=6) | Cohort 2 QBW276 (N=6) | Placebo (N=4)
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Feeling cold (General disorders) | 0 | 1 | 0
Mucosal dryness (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 3 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT02566044/SAP_000.pdf
  • Study Protocol (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT02566044/Prot_001.pdf